CLINICAL TRIAL: NCT01381497
Title: Impact of Migraine on Work Productivity in Patients Treated With a Combination Product Containing Sumatriptan and Naproxen Sodium or Triptan Monotherapy
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 112617
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Last update posted 2012-08-27 (Estimated); Status verified 2012-08

CONDITIONS: Migraine Disorders
Keywords: presenteeism; migraine disorders; work productivity; triptan; sumatriptan and naproxen sodium; absenteeism
MeSH Terms: conditions — Migraine Disorders | interventions — Naproxen; sumatriptan-naproxen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Employed migraine sufferers: Diagnosed adult migraine sufferers who are employed at least 30 hours per week during a daytime shift
  Interventions: Drug: Combination therapy of sumatriptan and naproxen sodium (SumaRT/Nap); Drug: Triptan monotherapy

INTERVENTIONS:
Drug: Combination therapy of sumatriptan and naproxen sodium (SumaRT/Nap) — This is an observational study and patients were prescribed this medication before study start
  Other Names: Treximet®
Drug: Triptan monotherapy — This is an observational study and patients reported a previous triptan monotherapy prescription. Drugs of interested included naratriptan, sumatriptan, rizatriptan, frovatriptan, almotriptan, eletriptan, zolmitriptan
  Other Names: Zomig® is a registered trademark of AstraZeneca; Amerge® is a registered trademark of GlaxoSmithKline; Axert® is a registered trademark of Pharmacia; Frova® is a registered trademark of Elan Pharmaceuticals/UCB Pharma; Inc; Maxalt® is a registered trademark of Merck & Co; Imitrex® is a registered trademark of GlaxoSmithKline; Relpax® is a registered trademark of Pfizer

SUMMARY:
Migraine headaches lead to absenteeism and can restrict on-the-job productivity (presenteeism) for employed migraine sufferers. Effective migraine treatments should reduce migraine-associated productivity losses and return migraineurs to normal functioning within a few hours of treatment.

This study is an observational, multicenter, parallel-group study of employed patients who have been prescribed either a combination product containing sumatriptan and naproxen sodium (SumaRT/Nap) or oral triptan monotherapy to treat acute migraine attacks. The study will report results from 4 migraine attacks per patient. Eligible migraine attacks will be defined as those preceded by a 24-hour, headache-free period with onset between 2 hours prior to the start of and 4 hours before the end of a scheduled work shift. Data will be collected at time of treatment and hourly until the end of the attack or the end of the workday. To estimate baseline productivity, data will be collected from 50 randomly selected subjects during a migraine-free workday.

The primary objective of this study is to compare migraine-related, work productivity losses (absenteeism and presenteeism) reported by patients treated with SumaRT/Nap to losses reported by patients treated with triptan monotherapy. The null hypothesis is that no difference will be observed between the number of hours of productivity lost for patients who treat workday migraine attacks with SumaRT/Nap and patients who treat migraine attacks with an oral triptan alone. The alternative hypotheses are that patients in either treatment group experience significantly fewer hours of lost productivity associated with migraine compared to patients in the other treatment group.

The secondary objectives of this study are to measure the time between treatment and return to patient-reported, normal functioning; to evaluate rescue medication use after initial treatment; to measure total productivity loss following treatment at hourly time points; and to estimate the probability of absenteeism when a migraine begins before or during the workday. The null hypotheses for the secondary endpoints are that no differences will be observed between the results reported by patients treating with SumaRT/Nap and patients treating with triptan monotherapy. The alternative hypotheses are that either treatment is superior to the other for each endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65
* Currently treating migraine attacks with SumaRT/Nap or oral triptan monotherapy
* Have a diagnosis of migraine with or without aura (2004 International Classification of Headache Disorders (ICHD)-II criteria)
* Have had at least 2 but not more than 8 migraine attacks per month in the previous 2 months
* Score 56 or higher on the Headache Impact Test 6 (HIT-6)
* Be actively employeed for at least 30 hours per week and working a day time shift (beginning between 6 and 11 AM)
* Have experienced and treated a disabling migraine in the work place during the month prior to screening
* Be willing to treat a mild, moderate, or severe migraine in the work place with usual medication (SumaRT/Nap or oral triptan alone)
* Be willing to adhere to protocol requirements including, but not limited to, hourly phone calls from the Interactive Voice-Activated Recording System (IVRS) and clinic visits
* Have an active cell phone with a plan that has sufficient monthly minutes during the study period to collect data via IVRS and be willing to provide their cell phone number to the study team
* Consent to phone the IVRS at the onset of a migraine attack during or prior to the workday and receive up to 8 phone calls (1 to 2 minutes each) during the workday.
* Be able to distinguish migraine attacks from other headache types
* Be able to hear, understand, and verbally answer questions from the IVRS in English
* Be willing and able to give written informed consent to participate in the study
* Female subjects of childbearing potential must use a reliable method of birth control as agreed upon by their investigator or male partner who is physiologically or surgically sterile. Any subject taking oral contraceptives must be on a stable regimen for at least two months prior to screening.

Exclusion Criteria:

* Subject often treats migraine attacks with a combination of a single entity triptan and any other medication
* Has 15 or more headache days per month in total, retinal (ICH-II 1.4), basilar (ICHD-II 1.26) or hemiplegic migraine (ICHD-II 1.25), or secondary headaches
* Has a HIT-6 score below 56 at screening
* Works an evening or night shift or works from home
* Has hypersensitivity, allergy, intolerance, or contraindication to any triptan or non-steriodal anti-inflammatory (NSAID) drug including aspirin and all sumatriptan and naproxen preparations.
* Has nasal polyps or asthma
* Is currently taking, or has taken in the 2 weeks prior to screening, a migraine prophylactic medication containing methylsergide or dihydroergotamine; or is takign a medication that is not stablized (i.e. change of dose within the previous two months) for intermittant migraine prophylaxis or for a co-morbid condition that is not stablized
* Has a recent history of regular use of opioids or barbituates for treatment of their migraine headache and/or other non-migraine pain. Regular use is defined as an average of 4 days per month during any month over the last 3 months
* Has taken or plans to take a monoamine oxidase (MAOI) inhibitor including herbal preparations containing St. John's Wort (Hypericum perforatum) anytime within the 2 weeks prior to screening through 2 weeks post final study treatment
* Is pregnant, actively trying to become pregnant, or breast feeding
* Has evidence of alcohol or substance abuse within the last year or any concurrent medical or psychiatric condition which, in the investigator's judgement, will likely interfere with the study conduct, subject cooperation, or evaluation and interpretation of the study results, or which otherwise contraindicates participation in this clinical trial
* Has participated in an investigational drug trial within the previous 4 weeks or plans to participate in another study at any time during this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult males and females aged 18 to 65 with a diagnosis of migraine disorder who are employed and scheduled to work at least 30 hours per week during a day time shift. Patients must be treating migraines with either a combination therapy of sumatriptan and naproxen sodium (SumaRT/Nap) or oral triptan monotherapy as prescribed prior to study start. Patients will be recruited from up to 30 investigative sites.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2010-03; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Total Lost Productivity (absenteeism and presenteeism) measured by Lost Time Equivalents | Four qualifying migraine attacks must occur within 16 weeks of enrollment. Data collection begins at time of treatment and continues in hourly intervals until the end of the migraine attack or the end of the workday.
  Lost Time Equivalents = hours missed from work + [(100% - % effectiveness while working with symptoms)/100 x hours working with symptoms].

SECONDARY OUTCOMES:
Percentage of patients returning to normal functioning as measured by the Clinical Disability Questionnaire (CDQ) | At time of treatment for a qualifying attack and at hourly intervals post treatment until end of migraine attack or end of workday
  The CDQ uses one question to assess ability to perform normal or usual activities. Responses are recorded on a 5-point scale, where 1 is "normal/not impaired", 2 is "mildly impaired", 3 is "moderately impaired", 4 is "severely impaired", and 5 is '"required bedrest". Normal functioning is considered a score of "1"
Rescue medication | Rescue medication is prohibited within 2 hours of study treatment administration. Rescue medication use is measured between 2 and 4 hours post treatment
  For patients who need pain relief in addition to the study treatment, rescue medication is allowed and measured. Type of rescue medication will be allowed at the discretion of the investigator and within the guidelines of the package insert for the study medication
Number of missed work hours and presenteeism hours lost following treatment measured in hours | At time of treatment for a qualifying attack and hourly intervals post treatment until end of migraine attack or end of workday
  Measured as per the primary endpoint and reported hourly
Probability of absenteeism during a morning migraine attack | At time of treatment for a qualifying attack and hourly intervals post treatment until end of migraine attack or end of workday
  A subgroup analysis will be conducted to provide information about the probability that patients will be absent if the migraine onset occurs in the morning

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline